CLINICAL TRIAL: NCT05458271
Title: Cross-linked Volume-stable Collagen Matrix Versus Connective Tissue Graft for Soft Tissue Augmentation At Implant Site. a Comparative, Multicentre Randomized Clinical Trial
Brief Title: Cross-linked Volume-stable Collagen Matrix Versus Connective Tissue Graft At Implant Site.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Dr. Francesco Cairo, Prof., University of Florence
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VCMX vs CTG
Record Dates: First submitted 2022-07-05; First posted 2022-07-14 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Edentulous Alveolar Ridge Atrophy; Soft Tissue Augmentation At Dental Implants

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Examiners will be blinded throughout all experimental procedures for all measurements.
  Operators will be blinded until they will raise the flap and screw the healing abutment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VCMX (Experimental): All patients will be treated by scaling/root planing to obtain infection control if needed. In addition, patients will receive oral hygiene instructions.
  The test group will be treated with add of VCMX. Following the local anesthesia, a split thickness flap will be raised-up to uncover the implant screw. Care will be taken to preserve pre-existing KT amount. A mesio-distal and apical partial thickness dissection will be performed to release residual muscle tension and allow the passive apical displacement of the flap. The randomisation envelope will be then opened. In test group the VCMX will be gently shaped and secured under the flap with suture. Care will be applied to completely cover the xenograft.
  Interventions: Device: VCMX
- CTG (Active Comparator): The control group patients will be treated by flap surgery with add of CTG. In the control group (APF) a CTG harvested from palate will be secured under the flap with suture.
  Interventions: Procedure: CTG

INTERVENTIONS:
Device: VCMX — A flap will be raised and VCMX will be placed in order to increase the soft tissue volume
  Arms: VCMX
Procedure: CTG — A flap will be raised and a CTG will be harvested from the palate and placed in order to increase the soft tissue volume
  Arms: CTG

SUMMARY:
Recent data suggested that an adequate volume of Keratinized Tissue (KT) around dental implant is a key factor to obtain aesthetic outcomes and to support easy long-term maintenance.

The aim of this RCT is to test the volume-stable collagen matrix (VCMX) vs the Connective Tissue Graft (CTG) for peri-implant soft tissue augmentation during implant uncovering.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* No systemic diseases or pregnancy.
* Self-reported smoking ≤10 cigarettes/day.
* No probing depths ≥5 mm
* Full-mouth plaque score (FMPS) and full-mouth bleeding score (FMBS) ≤15% (measured at four sites per tooth).
* Single dental implant with a scheduled for soft tissue augmentation procedure at the time of uncovering.
* Need of soft tissue augmentation for aesthetic purpose and/or functional reasons
* No previous soft tissue augmentation procedure at experimental site.

Exclusion Criteria:

* General contraindications for dental and/or surgical treatments
* Concurrent or previous immunosuppressant, bisphosphonate or high dose corticosteroid therapy
* Inflammatory and autoimmune disease of oral cavity
* History of myeloma, respiratory tract cancer, breast cancer, prostate cancer or kidney cancer requiring chemotherapy or radiotherapy within the past five years
* Radiotherapy of head area
* Disease or condition affecting connective tissue metabolism (e.g. disease of arteries in the operating zone, bone metabolic diseases, alcohol abuse, treatment with anticoagulants)
* Any systemic diseases that affect bone metabolism (e.g thyroid dysfunction, autoimmune disease)
* Untreated acute periodontal disease
* Patients who smoke more than 10 cigarettes/day will be excluded from the study
* Diabetes
* Allergy to the collagen
* Pregnant or lactating women
* Women of child bearing age, not using a highly effective method of birth control
* Participation in an investigational device, drug or biologic study within the last 24 weeks prior to the study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-07-31 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
GT | Immediately After Surgery
  Changes in the gingival thickness (in mm) measured 1.0 mm coronal to the MGJ using an injection needle, perpendicular to the tissue surface, with a silicon stop over the gingival surface.
GT | 1 week After surgery
  Changes in the gingival thickness (in mm) measured 1.0 mm coronal to the MGJ using an injection needle, perpendicular to the tissue surface, with a silicon stop over the gingival surface.
GT | 2 weeks After surgery
  Changes in the gingival thickness (in mm) measured 1.0 mm coronal to the MGJ using an injection needle, perpendicular to the tissue surface, with a silicon stop over the gingival surface.
GT | 4 weeks After surgery
  Changes in the gingival thickness (in mm) measured 1.0 mm coronal to the MGJ using an injection needle, perpendicular to the tissue surface, with a silicon stop over the gingival surface.
GT | 3 months After surgery
  Changes in the gingival thickness (in mm) measured 1.0 mm coronal to the MGJ using an injection needle, perpendicular to the tissue surface, with a silicon stop over the gingival surface.
GT | 6 months after surgery
  Changes in the gingival thickness (in mm) measured 1.0 mm coronal to the MGJ using an injection needle, perpendicular to the tissue surface, with a silicon stop over the gingival surface.
GT | 12 months after surgery
  Changes in the gingival thickness (in mm) measured 1.0 mm coronal to the MGJ using an injection needle, perpendicular to the tissue surface, with a silicon stop over the gingival surface.

SECONDARY OUTCOMES:
PROMs | Immediately After Surgery
  After explanation of the post-operative instructions patients will be given an evaluation questionnaire. Patient discomfort during procedure (from 0 to 10) and the overall judgment about the self-perception of procedure difficulty will be assed using a Visual Analogue Scale (VAS- (from 0 to 100))
PROMs | 1 week After surgery
  After explanation of the post-operative instructions patients will be given an evaluation questionnaire. Patient discomfort during procedure (from 0 to 10) and the overall judgment about the self-perception of procedure difficulty will be assed using a Visual Analogue Scale (VAS- (from 0 to 100)
PROMs | 2 weeks After surgery
  After explanation of the post-operative instructions patients will be given an evaluation questionnaire. Patient discomfort during procedure (from 0 to 10) and the overall judgment about the self-perception of procedure difficulty will be assed using a Visual Analogue Scale (VAS- (from 0 to 100)
PROMs | 4 weeks After surgery
  After explanation of the post-operative instructions patients will be given an evaluation questionnaire. Patient discomfort during procedure (from 0 to 10) and the overall judgment about the self-perception of procedure difficulty will be assed using a Visual Analogue Scale (VAS- (from 0 to 100)
PROMs | 3 months After surgery
  After explanation of the post-operative instructions patients will be given an evaluation questionnaire. Patient discomfort during procedure (from 0 to 10) and the overall judgment about the self-perception of procedure difficulty will be assed using a Visual Analogue Scale (VAS- (from 0 to 100)
PROMs | 6 months after surgery
  After explanation of the post-operative instructions patients will be given an evaluation questionnaire. Patient discomfort during procedure (from 0 to 10) and the overall judgment about the self-perception of procedure difficulty will be assed using a Visual Analogue Scale (VAS- (from 0 to 100)
PROMs | 12 months after surgery
  After explanation of the post-operative instructions patients will be given an evaluation questionnaire. Patient discomfort during procedure (from 0 to 10) and the overall judgment about the self-perception of procedure difficulty will be assed using a Visual Analogue Scale (VAS- (from 0 to 100)
KT | At Baseline
  The distance between muco-gingival junction, in mm, (MGJ) to the most coronal point of the ridge using a periodontal probe
KT | 1 week After surgery
  The distance between muco-gingival junction, in mm, (MGJ) to the most coronal point of the ridge using a periodontal probe
KT | 2 weeks After surgery
  The distance between muco-gingival junction, in mm, (MGJ) to the most coronal point of the ridge using a periodontal probe
KT | 4 weeks After surgery
  The distance between muco-gingival junction, in mm, (MGJ) to the most coronal point of the ridge using a periodontal probe
KT | 3 months After surgery
  The distance between muco-gingival junction, in mm, (MGJ) to the most coronal point of the ridge using a periodontal probe
KT | 6 months after surgery
  The distance between muco-gingival junction, in mm, (MGJ) to the most coronal point of the ridge using a periodontal probe
KT | 12 months after surgery
  The distance between muco-gingival junction, in mm, (MGJ) to the most coronal point of the ridge using a periodontal probe

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi di Firenze, Florence, FI, Italy

IPD SHARING:
Plan to Share IPD: Undecided